CLINICAL TRIAL: NCT01260272
Title: A Randomized, Unblinded, Single Research Site, Comparator Study of Raisins Versus Alternative Snacks on Cardiovascular Risk Factors In Generally Healthy Subjects
Brief Title: Study of Raisins Versus Alternative Snacks on Cardiovascular Risk Factors In Generally Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisville Metabolic and Atherosclerosis Research Center (Other)
Collaborators: California Raisin Marketing Board (Other)
Responsible Party: Principal Investigator, Harold E. Bays, Principal Investigator, Louisville Metabolic and Atherosclerosis Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Results first posted 2012-11-01 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Cardiovascular Risk Factors
Keywords: Cardiovascular; Risk Factors; Cardiovascular Disease; Glucose; Blood Pressure; BMI; Weight; Waist Circumference
MeSH Terms: conditions — Cardiovascular Diseases; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alternative Snack Group (Active Comparator): This group will receive 100 calorie alternative snack packs to consume three times a day with meals. Any prepackaged commercial snack is permitted as an alternative comparator snack, as long as it is 100 kcal/serving, does not contain raisins, does not contain solely fruits, and/or does not contain solely vegetables
  Interventions: Other: Alternative Snack Comparator
- Raisin Group (Experimental): This group will receive raisins to consume three times a day with meals
  Interventions: Other: Raisins

INTERVENTIONS:
Other: Alternative Snack Comparator — Any prepackaged commercial snack is permitted as an alternative comparator snack, as long as it is 100 kcal/serving, does not contain raisins, does not contain solely fruits, and/or does not contain solely vegetables. Preferred comparator snack examples include: Keebler® Cheez-It® Crackers, Fudge Shoppe ® Grasshopper® Cookies, Fudge Shoppe ® Mini Fudge Stripes ™ Cookies, Nabisco Chips Ahoy! Baked Chocolate Chip Snacks, Honey Maid Cinnamon Roll Thin Crisps, Lorna Doone Baked Shortbread Cookie Crisps, Oreo Baked Chocolate Wafer Snacks, Pepperidge Farm® Goldfish® Baked Snack Crackers
  Arms: Alternative Snack Group
Other: Raisins — Raisins are dry grape fruits that may be eaten raw, or used in cooking, baking, and brewing. Raisins are mostly composed of carbohydrates (mostly fructose). They are also high in fiber and antioxidants, relatively high in potassium, and low in sodium.
  Arms: Raisin Group

SUMMARY:
This trial compared the effects of raisin intake on cardiovascular risk factors compared to common, commercially available, alternative snacks. These cardiovascular risk factors include glucose, blood pressure, lipid levels, body weight, and waist circumference.

ELIGIBILITY:
Inclusion Criteria:

1. Are generally healthy men and women older than 18 years of age.
2. Are willing and able to undergo the informed consent process.
3. Have body mass index (BMI) from 25.0 to 34.9 kg/m².
4. Have one or more fasting plasma or serum glucose values of 90-150 mg/dl documented within 4 weeks of the initial study visit, or upon safety lab evaluation at the initial study visit.
5. Have blood pressure > 120 mmHg systolic or > 80 mmHg diastolic.
6. Are willing to notify the research staff of any change in their medical health & concomitant medications/supplements during the course of the clinical trial.

Exclusion Criteria:

1. Intolerance, dislike, or unwillingness to consume raisins or any of the comparator snacks and affiliated ingredients.
2. History of > one "food allergy."
3. Weight loss of > 5 pounds in last 2 months
4. Prior diagnosis of diabetes mellitus or currently taking diabetes mellitus drugs (including drugs such as metformin and colesevelam HCl, even if not being taken for diabetes mellitus). Subjects with prior history of gestational diabetes mellitus are eligible, as long as they no longer have diabetes mellitus, and are no longer taking medications for diabetes mellitus.
5. Blood pressure >160 mmHg systolic or >100 mmHg diastolic.
6. Fasting serum lipoprotein values of: LDL-cholesterol, >160 mg/dl or triglycerides, >500 mg/dl.
7. Creatinine level > 1.5 times the upper range of normal.
8. Potassium level above the upper range of normal (one repeat lab would be permitted if the initial elevated potassium level is thought possibly due to laboratory error)
9. Use of any medication or supplement to treat diabetes mellitus or blood glucose management at, or within 2 months prior to initial study entry.
10. Initiation or change of any antihypertensive medication within the two months prior to initial study entry. Subjects would be eligible if on stable dose of one or two antihypertensive medications that is/are to be maintained at constant dose throughout the study.
11. Initiation or change of any lipid-altering drug within the two months prior to initial study entry. Subjects would be eligible if on stable dose of one or two lipid-altering drugs that is/are to be maintained at constant dose throughout the study.
12. Is pregnant, breastfeeding or plans to become pregnant during the next three months.
13. Is an employee or immediate family member of the research staff.
14. Donated blood within 2 months prior to study entry, or plans to donate blood during the course of this study.
15. Use of systemic corticosteroids (intravenous, subcutaneous, intra-articular). Inhaled and intranasal corticosteroids are permitted.
16. Use of antiobesity/weight maintenance drug therapies at initial study visit, or within 2 months of the initial study visit.
17. Known medical history of clinical significance, or any other conditions that would present unacceptable risk to study subject, compromise the acquisition or interpretation of study data, or otherwise interfere with the study subject's participation in the study as per discretion of the Principal Investigator.
18. History of severe or uncontrolled depression based on Principal Investigator.
19. Known laboratory abnormalities prior to randomization which Principal Investigator deems may pose an unacceptable risk, compromise acquisition or interpretation of study data, or otherwise interfere with the study subject's participation in the study.
20. Major surgical procedure within 30 days prior to visit #1 (i.e. day of signing of the informed consent document), or current plans to have a major surgical procedure during study participation or 30 days following completion of all study related procedures.
21. History of gastrointestinal malabsorption (e.g. uncontrolled crohn's disease, etc.) or history of a gastric bypass or other diversional bariatric surgery. Gastric banding procedure is also exclusionary if adjusted within 30 days prior to visit #1 (i.e. day of signing the informed consent document), or a reasonable chance of having a gastric banding adjustment during the course of the study.
22. History of ongoing malignancy. Malignancy that has been successfully treated, with no evidence of persistence or recurrence of the malignancy within 5 years of visit #1 (i.e. day of signing the informed consent document) or basal carcinoma of the skin and "in situ" cancer of the cervix successfully treated 30 days prior to visit #1 are acceptable.
23. History of organ transplant.
24. History of drug (licit or illicit) or alcohol abuse/addiction within 5 years of visit #1 (i.e. day of signing the informed consent document).
25. Consumes more than 2 units of alcohol per day. A unit of alcohol is defined as a 12 ounce (350 ml) beer, 5 ounce (150 ml) wine, or 1.5 ounce (45 ml) of 80-proof alcohol for mixed drinks.
26. Known positive testing for hepatitis B surface antigen, hepatitis C antibody, active hepatitis A immunoglobulin M, or human immunodeficiency virus.
27. Anticipation of a significant change in job, job duties, or job work hours, which might impair their ability and willingness to undergo study-related procedures under the timelines specified by protocol, and otherwise impede their completion of the study.
28. Anticipation of or a reasonable likelihood of moving away from the research site, wherein such a move might impair their ability and willingness to undergo study-related procedures within the timelines specified by protocol, or otherwise impede their completion of the study.
29. Anticipation of or a reasonable likelihood of vacations or other times away from home which might impair their ability and willingness to undergo study-related procedures within the timelines specified by the study protocol, or otherwise impede their completion of the study.
30. Planned or anticipated major changes in lifestyle health practices, unless allowed by study protocol. Therapeutic Lifestyle Changes counseling will take place at randomization.
31. Treatment with an investigational product or an investigational device within 30 days prior to visit #1 (i.e. day of signing the informed consent document) and have no plans to potentially start any investigational product or use an investigational device during or 30 days after the study subject completes all study related procedures.
32. Reasonable life-expectancy of less than 2 years.
33. Any other reason, if in the opinion of the Investigator, the individual study subject is not appropriate, or suitable for participation in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold E. Bays, MD, Principal Investigator — Louisville Metabolic and Atherosclerosis Research Center
Locations (1):
- Louisville Metabolic and Atherosclerosis Research Center, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Anderson JW, Weiter KM, Christian AL, Ritchey MB, Bays HE. Raisins compared with other snack effects on glycemia and blood pressure: a randomized, controlled trial. Postgrad Med. 2014 Jan;126(1):37-43. doi: 10.3810/pgm.2014.01.2723. PMID 24393750

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study started around Dec 2010 and ended around April 2011. Subjects were selected from the PI's contact database and from advertisements
Pre-assignment Details: Subjects completed a 2-4 week screening period, during which labs and medical records were reviewed to verify eligibility
Groups:
- Alternative Snack Group: This group will receive 100 calorie alternative snack packs to consume three times a day with meals. Any prepackaged commercial snack is permitted as an alternative comparator snack, as long as it is 100 kcal/serving, does not contain raisins, does not contain solely fruits, and/or does not contain solely vegetables
  Alternative Snack Comparator : Any prepackaged commercial snack is permitted as an alternative comparator snack, as long as it is 100 kcal/serving, does not contain raisins, does not contain solely fruits, and/or does not contain solely vegetables. Preferred comparator snack examples include: Keebler® Cheez-It® Crackers, Fudge Shoppe ® Grasshopper® Cookies, Fudge Shoppe ® Mini Fudge Stripes ™ Cookies, Nabisco Chips Ahoy! Baked Chocolate Chip Snacks, Honey Maid Cinnamon Roll Thin Crisps, Lorna Doone Baked Shortbread Cookie Crisps, Oreo Baked Chocolate Wafer Snacks, Pepperidge Farm® Goldfish® Baked Snack Crackers
- Raisin Group: This group will receive raisins to consume three times a day with meals
  Raisins : Raisins are dry grape fruits that may be eaten raw, or used in cooking, baking, and brewing. Raisins are mostly composed of carbohydrates (mostly fructose). They are also high in fiber and antioxidants, relatively high in potassium, and low in sodium.
Period: Overall Study
Arm/Group | Alternative Snack Group | Raisin Group
Started | 17 | 32
Completed | 15 | 30
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alternative Snack Group | Raisin Group | Total
Number analyzed (Participants) | 17 | 32 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 20 | 33
  >=65 years | 4 | 12 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (1) | 60.3 (1) | 60.57 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 19 | 25
  Male | 11 | 13 | 24
Region of Enrollment [Number; unit: participants]
  United States | 17 | 32 | 49

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Postprandial Glucose Levels
Description: Raisins compared with snacks: percent change in postprandial glucose levels from baseline to week 12
Time Frame: 12 weeks
Population: Total # for analysis may not equal the randomized #. A last observation carried forward approach was utilized for those who did not complete the study, and who had at least 1 post treatment value. Subjects without at least 1 post treatment values were not included in the analysis. The analysis # was also adjusted by excluding defined outliers.
Measure: Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Alternative Snack Group | Raisin Group
Number analyzed (Participants) | 15 | 28
Percent change from baseline | 6.34 (7.4) | -9.83 (3.64)
Statistical Analysis 1: Comparison: Alternative Snack Group vs Raisin Group; Test type: Superiority or Other; p = 0.033, t-test, 2 sided — Apriori threshold for statistical significance was <=0.05

2. Secondary Outcome: Change in Systolic Blood Pressure
Description: Raisin versus snacks: change in systolic blood pressure from baseline to week 12
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Alternative Snack Group | Raisin Group
Number analyzed (Participants) | 14 | 30
mmHg | 1.71 (2.43) | -4.83 (1.86)
Statistical Analysis 1: Comparison: Alternative Snack Group vs Raisin Group; Test type: Superiority or Other; p = 0.0468, t-test, 2 sided — Apriori threshold for statistical significance was <=0.05

3. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Raisin versus snacks: change in diastolic blood pressure from baseline to week 12
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Alternative Snack Group | Raisin Group
Number analyzed (Participants) | 15 | 31
mmHg | -1.87 (2.14) | -5.16 (1.48)
Statistical Analysis 1: Comparison: Alternative Snack Group vs Raisin Group; Test type: Superiority or Other; p = 0.2114, t-test, 2 sided — Apriori threshold for statistical significance was <=0.05

4. Secondary Outcome: Change in Hemoglobin A1c
Description: Raisin versus snacks: change in hemoglobin A1c from baseline to week 12
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Alternative Snack Group | Raisin Group
Number analyzed (Participants) | 14 | 30
Percent change from baseline | -.04 (0.04) | -0.12 (0.04)
Statistical Analysis 1: Comparison: Alternative Snack Group vs Raisin Group; Test type: Superiority or Other; p = 0.1727, t-test, 2 sided — Apriori threshold for statistical significance was <=0.05

5. Primary Outcome: Percent Change in Fasting Glucose Levels
Description: Raisins versus snacks: percent change in fasting glucose levels from baseline to week 12
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | Alternative Snack Group | Raisin Group
Number analyzed (Participants) | 14 | 31
Percent change from baseline | 1.5 [-2.0 to 3.0] | 1.0 [-2.88 to 7.66]
Statistical Analysis 1: Comparison: Alternative Snack Group vs Raisin Group; Test type: Superiority or Other; p = 0.7498, Wilcoxon (Mann-Whitney) — Apriori threshold for statistical significance was <=0.05

6. Primary Outcome: Percent Change in Body Weight
Description: Raisin versus snacks: percent change in body weight from baseline to week 12
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Alternative Snack Group | Raisin Group
Number analyzed (Participants) | 14 | 31
Percent change from baseline | -0.67 (0.47) | 0.16 (0.44)
Statistical Analysis 1: Comparison: Alternative Snack Group vs Raisin Group; Test type: Superiority or Other; p = 0.2615, t-test, 2 sided — Apriori threshold for statistical significance was <=0.05

7. Secondary Outcome: Change in Waist Circumference
Description: Raisin versus snacks: change in waist circumference from baseline to week 12
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cm
Arm/Group | Alternative Snack Group | Raisin Group
Number analyzed (Participants) | 14 | 29
cm | -1.59 (0.52) | -2.02 (0.7)
Statistical Analysis 1: Comparison: Alternative Snack Group vs Raisin Group; Test type: Superiority or Other; p = 0.6915, t-test, 2 sided — Apriori threshold for statistical significance was <=0.05

8. Secondary Outcome: Change in High Density Lipoprotein Cholesterol Levels
Description: Raisin versus snacks: percent change in high density lipoprotein cholesterol levels from baseline to week 12
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Alternative Snack Group | Raisin Group
Number analyzed (Participants) | 13 | 30
Percent change from baseline | 0.62 (3.15) | -5.63 (2.08)
Statistical Analysis 1: Comparison: Alternative Snack Group vs Raisin Group; Test type: Superiority or Other; p = 0.1060, t-test, 2 sided — Apriori threshold for statistical significance was <=0.05

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the day the subject signed the Informed Consent Document, until 30 days after study completion.
Arm/Group | Alternative Snack Group | Raisin Group
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/32
Other Adverse Events (participants affected / at risk) | 5/17 | 20/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alternative Snack Group (N=17) | Raisin Group (N=32)
Decreased hunger (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Excess Gas (Gastrointestinal disorders) | 0 (0) | 1 (1)
Increased frequency of stools (Gastrointestinal disorders) | 0 (0) | 1 (1)
Indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Worsening hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Diabetes Mellitus (Endocrine disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Worsening heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Xerostomia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Allergic Rhinitis (General disorders) | 0 (0) | 1 (1)
Fluid retention (General disorders) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1)
Vertigo (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Elevated liver enzymes (Hepatobiliary disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Puncture wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — injury- not related to study
Posterior head pain related to trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left ankle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Strained muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Effusion to right elbow (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign uterine mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Intermittent cough (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chest congestion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Contusion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Brain hemorrhage (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a single research site pilot study, which would benefit from a larger study, or at least, a similar confirmatory study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes